CLINICAL TRIAL: NCT06500598
Title: Compassionate Use of Evinacumab
Status: Approved for marketing | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R1500-Evinacumab
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Homozygous Familial Hypercholesterolemia (HoFH); Severe Hypertriglyceridemia (HTG); Dysbetalipoproteinemia (DBL)
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipoproteinemia Type III | interventions — evinacumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Evinacumab
  Other Names: REGN1500; EVKEEZA®

SUMMARY:
Provide compassionate use of evinacumab

DETAILED DESCRIPTION:
Compassionate Use requests are only being considered in response to Individual Patient Investigational New Drug (IND) applications. Availability will depend on location.

Age Groups: Child, Adult, Older Adult